CLINICAL TRIAL: NCT00409435
Title: Double-Blind, Placebo-Controlled Study of Pyridostigmine in Postural Tachycardia Syndrome
Brief Title: A Study of Pyridostigmine in Postural Tachycardia Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Wolfgang Singer, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-002442; P01NS044233 (NIH)
Record Dates: First submitted 2006-12-06; First posted 2006-12-08 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Postural Tachycardia Syndrome
Keywords: Postural tachycardia syndrome (POTS)
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- pyridostigmine (Active Comparator): Active study drug
  Interventions: Drug: pyridostigmine
- Placebo (Placebo Comparator): Control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pyridostigmine — one 180 mg capsule per day for 3 days
  Arms: pyridostigmine
Drug: Placebo — one capsule per day for 3 days
  Arms: Placebo

SUMMARY:
This is a 3-day study comparing pyridostigmine versus placebo in the treatment of postural tachycardia syndrome (POTS). The researchers expect pyridostigmine to improve tachycardia and stabilize blood pressure.

DETAILED DESCRIPTION:
The study will be done at the outpatient General Clinical Research Center (GCRC) at Charlton 7 and will involve two visits. Visit 1 will take about 3 hours, and Visit 2 will occur 2 days after Visit 1 and will take about 2 hours.

You will be put in one of two groups by chance (as in the flip of a coin). One group will be taking placebo (an inactive substance), the other group 180 mg pyridostigmine in time release formulation. Both placebo and pyridostigmine will look identical and will be taken as one capsule per day for 3 days. Neither you nor the study doctor will know at the time of treatment whether the treatment being given is active or inactive. However, in case of an emergency, this information will be available.

For each of the two visits, the following tests and procedures will be performed:

* When you arrive at the GCRC, you will have a general medical and neurological examination and height and weight measurement.
* Questionnaires. You will be asked to answer a series of questions on your autonomic symptoms (such as rapid heart rate, feeling of tiredness, cold and sweaty hands) at each of your two visits. The questionnaire you will be given during your first visit should take approximately 30 minutes to complete. The questionnaire you will be given during your second visit should take approximately 10 minutes to complete.
* Autonomic Reflex Screen. An autonomic reflex screen will be done during each visit. This consists of the following:

  * Quantitative sudomotor axon reflex test (QSART): QSART is a routine clinical test that evaluates the response of the sweat gland to a drug, acetylcholine. One capsule is placed on your forearm and three on your leg and foot. The testing is done by passing a small electrical current, for 5 minutes, to activate the nerves that supply the sweat glands. You will feel a slight burning sensation.
  * Cardiovascular recordings: Blood pressure, heart rate, and other cardiovascular measurements will be studied by placing electrodes on the chest and a finger or wrist cuff for continuous blood pressure recordings.
  * Valsalva maneuver: This involves blowing very hard into a bugle (like blowing up a balloon) for 15 seconds.
  * Head-up tilt: Following a period of rest (at least 5 minutes), you will be tilted up to an angle of not more than 80 degrees and recordings will be made for up to 30 minutes. On Visit 1, one hour after you have taken the study medication, this test will be repeated. This test will be done only once on Visit 2.
  * Hormone level measurements: This will be done during each visit. An IV will be inserted into a vein in your arm from which approximately one teaspoon of blood will be drawn while you are lying down and one teaspoon after standing up. This will be repeated only on Visit 1, one hour after the study drug is given. A total of four teaspoons of blood will be drawn on Visit 1 and 2 teaspoons will be drawn on Visit 2.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of postural tachycardia syndrome using the following criteria:

* Orthostatic heart rate increment greater than or equal to 30 beats per minute (bpm) within 5 minutes of head-up tilt.
* Symptoms of orthostatic intolerance. These include weakness, lightheadedness, blurred vision, nausea, palpitations, and difficulty with concentration and thinking.

Both criteria must be fulfilled.

Exclusion Criteria:

* Pregnant or lactating women
* Presence of failure of other organ systems or systemic illness that could affect autonomic function or the patient's ability to cooperate with the study
* Hypothyroidism or hyperthyroidism
* Clinically significant coronary artery disease
* Medications that could interfere with autonomic testing
* Previous treatment with pyridostigmine for POTS. Patients must not have taken pyridostigmine in the past month

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-10; Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in orthostatic symptoms using Composite Autonomic Symptom Scale (COMPASS) change | 3 days

SECONDARY OUTCOMES:
Heart rate response to head-up tilt | 3 days
Plasma norepinephrine change | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Singer, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Dani M, Fedorowski A. Tackling POTS Needs More Than Just a Sympathetic Approach. Hypertension. 2024 Nov;81(11):2248-2250. doi: 10.1161/HYPERTENSIONAHA.124.23716. Epub 2024 Oct 16. No abstract available. PMID 39413203
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials